CLINICAL TRIAL: NCT04251663
Title: Examine the Roles of Complement C5a Receptors in Hidradenitis Suppurativa by ex Vivo Studies
Brief Title: Complement C5a Receptors in Hidradenitis Suppurativa
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kavita Sarin, Assistant Professor of Dermatology, Stanford University
Other Study IDs: 51335
Record Dates: First submitted 2019-07-18; First posted 2020-02-05 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HS subjects: Subjects with active HS disease, among which at least 5 will be treatment-naïve
- Healthy Controls: Healthy subjects

SUMMARY:
To study the role of C5a in Hidradenitis Suppurativa (HS). Complement C5a is a major chemotactic factor that stimulates neutrophil infiltration.

DETAILED DESCRIPTION:
Hidradenitis suppurativa is a debilitating chronic inflammatory follicular skin disease. The estimated prevalence of HS range between 1 and 4%, even though it has been an underdiagnosed disease until recently (Revuz J, 2009). In the acute stage, patients present with painful inflamed nodules (boils) and abscesses in the groin, buttocks and axillae. In a late stage sinus tract formation and scarring occurs. Treatment options include the antibiotics, anti-TNF and surgical methods (wide excisions and deroofing). However, most patients do not respond, or only respond partially or temporarily to treatments (von der Werth JM, 2001; Napolitano M, 2017; Nazary M, 2011; van der Zee HH, 2012).

The pathogenesis of HS is largely unknown, and possible causes include plugged apocrine gland or hair follicle, excessive sweating, androgen dysfunction and genetic disorders. Defective cytokine responses and the infiltration of a variety of immune cells suggest the autoinflammatory nature of the disease (Giamarellos-Bourboulis EJ, 2007; van der Zee HH; 2011; van der Zee HH, 2012), which is in line with the significant improvement seen in patients administered the tumor necrosis factor-a (TNF-a) blocker adalimumab (Kimball AB, 2016). Neutrophils have been identified in skin lesions and are considered to be the major cell type to produce pus. Complement C5a is a major chemotactic factor that stimulates neutrophil infiltration. The role of C5a has just recently started to be studied in HS. (Blok JL, 2016; Kanni T, 2018). An open label phase 2 study demonstrated that a 50% HS clinical response rate was achieved in up to 83% of patients receiving an C5a antibody (IFX-1, NCT 03001622). Thus, targeting the C5a signaling may represent a promising therapeutic strategy in HS.

Most of the C5a effects result from binding to the canonical complement 5a receptor 1, C5aR. However, there is a second C5a receptor, C5L2, whose roles are still controversial. Both pro- and anti-inflammatory properties have been proposed for C5L2. These contradictory results may be dependent on specific physiological or pathological conditions (Zhang T, 2017). ChemoCentryx has a series of potent and selective small molecule C5aR inhibitors (C5aRi) that are being developed for inflammatory diseases such as ANCA associated vasculitis, C3 glomerulopathy and HS. In this proposal, we will use these C5aRi to examine the differential effects of targeting C5aR.

Study Design

An ex vivo skin culture system will be utilized to examine the effects of C5aR inhibition on neutrophil activation/inflammatory activities. Four-millimeter (4mm) lesional and perilesional skin biopsies will be taken from skin excisions of 40 patients with known Hidradenitis Suppurativa. Surplus skin excision material from "deroofment" treatment of HS patients will be used. Peri-lesional and lesional biopsies will be collected for comparison. These samples will be delivered to ChemoCentryx for direct analysis or treatment with C5a and/or C5a inhibitors. Analysis will include but not limited to histological analysis, examining immune cell populations and surface markers, protein and gene expression levels of complement factors, cytokines and chemokines. Flow cytometry, immunohistochemistry, ELISA and other standard assays will be used for these analyses. These studies will extend the on-going studies with Dr. Kavita and colleagues, and will test the hypothesis that continued activation of neutrophils and other C5a-expressing leukocytes in the skin lesions of HS patients contribute to tissue damage.

We plan to collect plasma samples from 40 HS patients with active disease. All sample collection will follow a well-defined protocol, with a maximum of 30ml of blood collected. Samples will be immediately transported to ChemoCentryx for processing. Immune cell populations, expression levels of C5aR and other related factors, responses to ex vivo stimulations, and other characteristics of blood cells will be examined. Plasma and serum will be collected and analyzed for levels of complement factors, cytokines and chemokines. The plasma samples will also be used to stimulate immune cells purified from health donors. C5a and C5aR inhibitor will be used to determine the role of C5aR in these in vitro assays.

Participants will be consented and enrolled for a single initial study visit with collection of blood and/or skin tissue. Completion of this visit will be considered the end of the individual's participation in the study. Participants may, however, at the discretion of the principle investigator, be consented and enrolled again for a future study visit with collection of blood and/or skin tissue. Re-enrolled participants will retain their initial study code and collected specimens will be date and visit number labelled.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to sign consent and provide a blood sample
* Willing to provide 2 skin biopsies - lesional and perilesional
* Active HS disease or healthy volunteer

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The team will collect plasma and tissue samples from 40 HS patients with active disease, among which at least 5 will be treatment-naïve. Plasma from 10 healthy volunteers will be used as controls. The team will try to obtain blood and 2 skin biopsies (1 from a HS lesion, 1 from normal skin).
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
CD11b surface expression on neutrophils | Day 1 study visit (up to 2 hours)
  Relative expression of adhesion molecule (CD11b) on circulating neutrophils in HS patients determined by flow cytometry.
C5aR surface expression on neutrophils | Day 1 study visit (up to 2 hours)
  Relative expression of canonical complement 5a receptor (C5aR) on circulating neutrophils in HS patients determined by flow cytometry.

SECONDARY OUTCOMES:
Immune cell population profiling | Day 1 study visit (up to 2 hours)
  Immune cell population profile as measured by the percentage of circulating neutrophils, macrophage and T cells as determined by flow cytometry.
Measurement of cytokines | Day 1 study visit (up to 2 hours)
  Skin biopsies will be cultured ex vivo. Cytokine profile as measured by the level of cytokines in assay supernatant by multiplex ELISA: IL-1β, IL-6, TNF-α, IL-12, IL-23, IL-17A, IL-17F, IFN-γ.

OTHER OUTCOMES:
Complement factor analysis | Day 1 study visit (up to 2 hours)
  Complement factor (such as C1q, C4d, Bb, iC3b, C5b-9) will be analyzed by immunohistochemistry on biopsy samples (pending extra tissue availability after flow cytometry analysis)..

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Y Sarin, MD PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No